CLINICAL TRIAL: NCT05467683
Title: Carbon Dioxide (CO2) Reactivity as a Biomarker of Non-Response to Exposure-Based Therapy
Brief Title: CO2 Reactivity as a Biomarker of Non-Response to Exposure-Based Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Boston University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jasper A. Smits, Professor of Psychology, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001631; 1R01MH125951-01A1 (NIH); 1R01MH125949-01A1 (NIH)
Record Dates: First submitted 2022-06-27; First posted 2022-07-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Obsessive-Compulsive Disorder; Post Traumatic Stress Disorder; Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Stress Disorders, Post-Traumatic; Generalized Anxiety Disorder; Phobia, Social; Panic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Exposure-Based Therapy (EBT) (Other): All participants will receive a well-established psychological treatment.
  Interventions: Behavioral: Exposure-Based Therapy

INTERVENTIONS:
Behavioral: Exposure-Based Therapy — Treatment will consist of 12 one-hour sessions, delivered over the course of 12 weeks. EBT will be delivered by trained and experienced license-eligible clinicians. The study clinician will develop a personalized assessment and treatment plan for each patient. Consistent with contemporary models of EBT, exposure practice aims to help patients reestablish a sense of safety around feared cues. Hence, exposure exercises are planned to ensure violation of threat expectancies. That is, exposure practice is deemed appropriate and effective if it allows the patient to learn that what they feared would happen does not happen. Practice will occur across relevant contexts both within and outside the session (i.e., homework) and clinicians will guide patients in processing practice to facilitate the consolidation of safety learning. To achieve these ends, study clinicians will use the manual "Personalized Exposure Therapy: A Person-Centered Transdiagnostic Approach".

SUMMARY:
Anxiety-, obsessive-compulsive and trauma- and stressor-related disorders reflect a significant public health problem. This study is designed to evaluate the predictive power of a novel biomarker based on a CO2 challenge, thus addressing the central question "can this easy-to-administer assay aid clinicians in deciding whether or not to initiate exposure-based therapy?"

DETAILED DESCRIPTION:
Exposure-based therapy is an effective first-line treatment for anxiety-, obsessive-compulsive and trauma- and stressor-related disorders. However, many patients fail to respond or achieve remission with exposure-based therapy, resulting in prolonged suffering, loss of productivity, and poorly used resources. Making available a biomarker assay that can aid clinicians and patients in treatment selection has the potential to have considerable public health impact.

Basic research on fear extinction--a core mechanism of action of exposure-based therapy--may inform the development of a biomarker for the selection (yes/no) of exposure-based therapy. Growing evidence links orexin system activity to deficits in fear extinction. Our group has demonstrated that reactivity to CO2 challenge, which is a safe, affordable and easy-to-implement procedure, can serve as a proxy for orexin system activity and predicts fear extinction deficits in rodents.

Building upon this basic research, the goal for the proposed study is to validate CO2 reactivity as a biomarker of exposure-based therapy non-response. To this end, we will assess CO2 reactivity in 600 adults meeting for one or more fear- or anxiety-related disorders prior to providing open, state-of-the art, transdiagnostic exposure-based therapy. By incorporating CO2 reactivity into a multivariable model predicting treatment non-response that also includes reactivity to hyperventilation as well as a number of related and theoretically-relevant prognostic variables, we will establish the mechanistic specificity and the additive predictive value of the putative biomarker. By developing models independently within two study sites and predicting the other site's data, we will validate that the results are likely to generalize to future clinical samples.

The proposed study represents a necessary stage in translating basic research to strategies for treatment selection. The investigation addresses an important public health issue by testing an accessible clinical assessment strategy--informed by basic research--that may lead to a more effective treatment selection (personalized medicine) for patients with anxiety- and fear-related disorders and enhance our understanding of the mechanisms governing exposure-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* A primary DSM-5 diagnosis of panic disorder (with or without an agoraphobia diagnosis), social anxiety disorder, generalized anxiety disorder, obsessive-compulsive disorder, or post-traumatic stress disorder as assessed by the Structured Clinical Interview for the DSM-5 (SCID-5)
* A score of 8 or greater on the Overall Anxiety Severity and Impairment Scale (OASIS)
* Ages 18 to 70
* Willingness and ability to provide informed consent and comply with the requirements of the study protocol.
* Proficiency in English (because assessment instruments have only been validated in English)

Exclusion Criteria:

* A lifetime history of bipolar or psychotic disorders, substance use disorders (other than nicotine) or eating disorder in the past 6 months; serious cognitive impairment.
* Active suicidal ideation with at least some intent to act with or without specific plan (a rating of 4 for suicidal ideation on the Columbia-Suicide Severity Rating Scale) or suicidal behaviors (actual attempt, interrupted attempt, aborted or self-interrupted attempt, or preparatory acts or behavior) within the past 6 months.
* Medical conditions contraindicating CO2 inhalation or hyperventilation challenge (e.g., cardiac arrhythmia, cardiac failure, asthma, lung fibrosis, high blood pressure, epilepsy, or stroke).
* Pregnancy or lactation
* Ongoing psychotherapy directed toward the primary disorder.
* Pharmacological treatment started within 8 weeks prior to the screen (patients "stable" on their medication regimen will be included and their medication status will be included as a variable in the model)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Non-response to exposure-based therapy | Week 13 (post-treatment)
  Participants will be classified as non-responders if their Clinical Global Impression - Global Improvement (CGI-I) score is 3 or above OR if their Overall Anxiety Severity and Impairment Scale (OASIS) score has not improved by at least 4 points.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity of Illness (CGI-S) | Weekly for 14 weeks + follow-up after 24 weeks
  A 7 point widely used clinician rating scale for indexing the how mentally ill a patient is at the time using a 7 point scale ranging from 1(normal, not at all ill); 2 (borderline mentally ill); 3 (mildly ill); 4 (moderately ill); 5 (markedly ill); 6 (severely ill); 7(among the most extremely ill patients).
Overall Anxiety Severity and Impairment Scale (OASIS) | Weekly for 14 weeks + follow-up after 24 weeks
  The OASIS is a self-report rating scale that comprises five items to assess the frequency and severity of anxiety, avoidance, work/school/home interference, and social interference due to anxiety. Participants select among five different response options for each item, which are coded 0-4 and are summed to obtain a total score (0-20).
GAD-7 | Weekly for 14 weeks + follow-up after 24 weeks
  For participants with generalized anxiety disorder (GAD) as their primary DSM-V diagnosis, intended to assess the severity of participant symptoms. Ranged from 0 to 21, with higher scores indicating more severe distress and impairment.
Panic Disorder Severity Scale (PDSS) | Weekly for 14 weeks + follow-up after 24 weeks
  For participants with panic disorder (PD) as their primary DSM-V diagnosis, intended to assess the severity of participant symptoms. Ranged from 0 to 28, with higher scores indicating more severe distress and impairment.
Social Phobia Inventory (SPIN) | Weekly for 14 weeks + follow-up after 24 weeks
  For participants with social anxiety disorder (SAD) as their primary DSM-V diagnosis, intended to assess the severity of participant symptoms. Ranged from 0 to 68, with higher scores indicating more severe distress and impairment.
Dimensional Obsessive-Compulsive Scale (DOCS) | Weekly for 14 weeks + follow-up after 24 weeks
  For participants with obsessive compulsive disorder (OCD) as their primary DSM-V diagnosis, intended to assess the severity of participant symptoms. Ranged from 0 to 80, with higher scores indicating more severe distress and impairment.
PTSD Checklist for DSM-5 (PCL-5) | Weekly for 14 weeks + follow-up after 24 weeks
  For participants with post-traumatic stress disorder (PTSD) as their primary DSM-V diagnosis, intended to assess the severity of participant symptoms. Ranged from 0 to 80, with higher scores indicating more severe distress and impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Smits, Ph.D., Principal Investigator — The University of Texas at Austin; Michael Otto, Ph.D., Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Boston University, Boston, Massachusetts
  - The University of Texas at Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
In line with National Institute of Mental Health (NIMH) guidance, we will share de-identified data derived from this study via the National Data Archive (NDA), along with supporting documentation to enable efficient and appropriate use of the data. Data sharing is now a requirement for all NIMH-funded awards (NOT-MH-14-015). Consistent with the National Database for Clinical Trials related to Mental Illness (NDCT) guidelines, we will share data in a two-tiered approach. The first tier involves semi-annual uploading of descriptive and raw data while the study is ongoing, including data from standard assessments, standard clinical measures, demographic data, and raw behavioral data. The second tier includes analyzed data that result from publications. We will ensure that submitted data will conform to relevant data and terminology standards. Throughout our resource sharing plan, we will comply with NDCT guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Descriptive/raw data will be shared on a semi-annual basis (on or before January 15 and July 15, beginning six months after the award budget period has begun). Analyzed data will be submitted prior to publication/public dissemination (whether the findings are positive or negative) using the NDA Study feature that links data deposited in the NDA with publications/findings.
Access Criteria: We agree that data will be deposited and made available through NDA, and that these data will be shared with investigators working at an institution with a Federal Wide Assurance (FWA) and could be used for secondary study purposes. All submitted data (both descriptive/raw and analyzed data) will be made available for access by qualified members of the research community according to the provisions defined in the NIMH Data Repositories Data Access Agreement and Use Certification.
URL: https://nda.nih.gov/edit_collection.html?id=4334

REFERENCES:
- [Derived] Smits JAJ, Monfils MH, Otto MW, Telch MJ, Shumake J, Feinstein JS, Khalsa SS, Cobb AR, Parsons EM, Long LJ, McSpadden B, Johnson D, Greenberg A; Exposure Therapy Consortium. CO2 reactivity as a biomarker of exposure-based therapy non-response: study protocol. BMC Psychiatry. 2022 Dec 27;22(1):831. doi: 10.1186/s12888-022-04478-x. PMID 36575425